CLINICAL TRIAL: NCT00120822
Title: A Study of the Effect of Folic Acid Supplementation on the Anti-malarial Action of Sulfadoxine-pyrimethamine When Used for Intermittent Preventive Treatment in Gambian Primigravidae.
Brief Title: Folic Acid Supplementation in Gambian Primigravidae
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Department of State for Health and Social Welfare, The Gambia (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ITCRVG27a
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Malaria; Pregnancy; Folic acid; Sulfadoxine-pyrimethamine
MeSH Terms: conditions — Malaria | interventions — Folic Acid

INTERVENTIONS:
Drug: Folic acid

SUMMARY:
Supplementation with folic acid and iron is recommended for pregnant women in order to prevent them from developing anemia. In malaria endemic areas of Africa, the World Health Organization (WHO) now recommends that pregnant women should also be given sulfadoxine-pyrimethamine (SP) once a month after quickening to protect them against malaria which is especially harmful during pregnancy. However, folic acid is an antagonist of SP so there is a possibility that giving folic acid with SP could interfere with the ability of the latter to provide protection against malaria. To investigate this possibility Gambian primigravidae with malaria parasitemia have been given SP and folic acid at the same time or on separate occasions two weeks apart and the ability of SP to cure the malaria infection investigated.

DETAILED DESCRIPTION:
Objective

The objective of this study is to determine if administration of folic acid to pregnant women at the same time as sulfadoxine-pyrimethamine (SP) is given to prevent malaria interferes with the protective effect of the SP.

Study area

The study was carried out in 14 mother and child health (MCH) clinics situated on the north and south banks of the River Gambia near to the town of Farafenni in the centre of the country. In this area malaria is highly seasonal with an entomological inoculation rate of 10-50 infectious bites per year.

Study population

Primigravidae who attended one of the study clinics were reviewed to assess their eligibility to join the study. Entry criteria were - pregnancy > 15 weeks, haemoglobin (Hb) > 7g/dl, absence of any underlying serious disease, absence of a history of an adverse reaction to sulfonamide, residence in the study area and a willingness to be visited at home.

Study procedure

Eligible women were asked if they wished to join the trial and, if so, written, informed consent was obtained. An entry questionnaire was then completed and a finger-prick blood sample obtained for determination of Hb and preparation of two thick blood films. Provided the woman had a Hb >7g/dl, she was then given a study number and formally entered into the trial. Women were then individually randomised to receive SP and iron + folic acid ('early' folate group) or SP and iron ('late' folate group).

All women in the trial received three tablets of SP (25 mg pyrimethamine and 500 mg sulfadoxine) (Cosmos Pharmaceutical, Nairobi) given under observation. Women in the 'early' folic acid group then received a packet containing Fefol (500 ug of folic acid and 47 mg of ferrous sulfate) to be taken at home once per day for 14 days. Women in the 'late' folic acid group received packets containing oral iron (60 mg/day) alone to be taken daily for 14 days. At the day 14 follow-up they then received iron and folic acid so no woman was deprived of folic acid supplementation.

At the end of the 14 day period, women were visited at home and a repeat finger-prick blood sample obtained for determination of Hb and preparation of two thick blood films.

Haemoglobin was measured using a Haemocue and blood films were examined for malaria parasites after staining with Giemsa by two microscopists blind to the treatment code. If discrepant results were found, a third reading was done and the majority view accepted.

Trial end-point

The primary end-point for the trial was the prevalence of Plasmodium falciparum asexual parasitemia 14 days after treatment in women who were parasitemic on presentation. Parasite prevalence at day 14 irrespective of initial findings and mean Hb at day 14 were secondary end-points.

Sample size

It was assumed that 30% of women would be parasitemic on presentation and that the cure rate with SP in those who did not receive folic acid at the same time would be 97%. To have 90% power at the 5% level of significance to show a 10% reduction in the cure rate with SP when this is given with folic acid, 483 women were required for each arm of the trial.

Data Safety Monitoring Board (DSMB)

A DSMB was established to monitor the conduct of the trial and to approve the analytical plan prior to the breaking of the study code. The trial was conducted in line with the requirements of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Primigravid pregnancy > 15 weeks
* Residence in study area
* Informed consent

Exclusion Criteria:

* Any serious underlying illness.
* History of adverse reaction to sulfonamides

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-07; Study Completion 2004-01

PRIMARY OUTCOMES:
Clearance of malaria parasitemia in parasitemic pregnant women 14 days after treatment with sulfadoxine-pyrimethamine.

SECONDARY OUTCOMES:
The prevalence of malaria parasitemia 14 days after administration of a dose of sulfadoxine-pyrimethamine to pregnant women.
The mean haemoglobin 14 days after administration of a single dose of sulfadoxine-pyrimethamine to pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Greenwood, MD, Study Chair — London School of Hygiene and Tropical Medicine
Locations (1):
- Medical Research Council, Laboratories, Banjul, The Gambia